CLINICAL TRIAL: NCT06308835
Title: Prevalence and Risk Factors of Post Intensive Care Syndrome at 3 Months of an Intensive Care Unit Stay for a Neurological Disease
Brief Title: Prevalence and Risk Factor of Post-intensive Care Syndrome in Neuro-ICU
Acronym: STRESSréa
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231652
Record Dates: First submitted 2024-03-05; First posted 2024-03-13 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Post Intensive Care Syndrome
MeSH Terms: conditions — postintensive care syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaires — BREF(Batterie d'efficience Frontale), SDMT (Symbol Digit Modalities Test), TMT (Trail making test), Empans verbaux et BNT (Boston naming Test)

SUMMARY:
Post-intensive care syndrome (PICS) is the set of disabling symptoms that can appear or worsen following a stay in intensive care. These symptoms are physical, cognitive, or psychiatric. The onset and persistence of these symptoms have a major impact on patients' quality of life, their autonomy, and their social and professional reintegration. patients with neurological diseases are frequently excluded from studies due to difficulties for the non-specialist resuscitator to perform the neurological examination and assess whether the symptoms of RPS are secondary to brain damage or complications inherent in resuscitation.The aim of this study is to evaluate the incidence and characteristics of PICS in patients with neurological diseases, at ICU discharge and 3 months after, and to identify the risk factors for developing it.

DETAILED DESCRIPTION:
"Post-intensive care syndrome (PICS) is defined as a new or worsening impairment in physical, cognitive or mental health status arising and persisting after a stay in intensive care unit (ICU) . The onset and persistence of these symptoms have a major impact on patients' quality of life, their autonomy, and their social and professional reintegration. PICS is very common, and more than half of ICU adult patients experience such impairments.

Recent French guidelines about PICS have been published and implemented to raise awareness among clinicians and patients about diagnosis and management of PICS .

A systematic ICU follow-up consultation by trained practitioners allows the diagnosis of PICS, and the implementation of appropriate curative measures to minimize sequelae and improve outcomes . This consultation is increasingly recommended by learned societies.

Incidence and risk factors of PICS is poorly known in patients with neurological diseases, because they are frequently excluded from PICS studies due to difficulties to assess whether the symptoms are disease-related or directly associated with the experience of a critical illness. A better knowledge of follow up of these patients is necessary to identify if some neurocognitive sequelae may be preventable or treatable.

The aim of this study is to evaluate the incidence and characteristics of PICS in patients with neurological diseases, at ICU discharge and 3 months after, and to identify the risk factors for developing it.

The investigators wish to conduct a bi-centric prospective study, in two neurological ICU in Paris (AP-HP Sorbonne université - Pitié Salpetrière hospital and Paris Cité -Saint Anne Hospital). The study will last one year.

It will included adults patients hospitalized >24h in neuro-ICU for a neurological disease affecting the central nervous system (status epilepticus, encephalitis, subarachnoid haemorrhage…) or the peripheral nervous system (myasthenia gravis crisis, Guillain-Barre syndrome…) ; and having received ICU lifesaving treatments (mechanical ventilation; sedation; plasmapheresis, renal replacement therapy, catecholamine).

Were excluded pregnant women, patients with pre-existing neurodegenerative disease or pre-existing severe psychiatric illness, and patients whose neurological or psychiatric history were not known prior to ICU. Patients with blindness, deafness, inability to speak French, active substance abuse, homelessness, or who lived > 100 kilometers from the enrolling center.

Patients will be recruited at the end of the ICU stay, patient's non-opposition will be collected. If the patient is unable to consent, the non-opposition of the person of trust will be collected.

As close as possible to the ICU discharge, a neurological examination, a MRC score, a MOCA scale, and a HADS scale will be performed.

The ICU-follow up visit will be planned 3 months +- 30 days from the ICU discharge and will include:

* An interview conducted by a trained neuro-intensivist with assessment of neurological symptoms and autonomy assessed by the Glasgow Outcome Scale extended (GOS-e), and the modified Rankin Scale (mRS), of psychiatric symptoms with self-reported questionnaires: Hospital Anxiety and Depression Scale (HADS) and the impact of event scale (IES-R).
* A physical assessement by a physiotherapist including a Medical research coucil score (MRC)
* A neuropsychological assessement by a neuropsychologist including a Montreal Cognitive Assessment (MOCA), batterie d'efficience frontale (BREF), Symbol Digit Modalities Test (SDMT), Trail Making Test (TMT), Empans verbaux, Boston naming Test (BNT)

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient with > 24h stay in intensive care unit
* 2.Patients with a neurological disease affecting the central or peripheral nervous system, which is the reason for their hospitalization in intensive care.
* 3. Patients who have received organ replacement or invasive therapy in the ICU (invasive or non-invasive ventilation, extra-renal purification, plasmapheresis, ventricular bypass, catecholamines).
* 4. Non-opposition of the patient or of the trusted support person, or of a family member or close friend if the patient is unable to express non-opposition.

Exclusion Criteria:

* 1. Minors, protected adults and pregnant women
* 2. Advanced neurodegenerative disease pre-existing prior to ICU admission
* 3. Severe psychotic disorders pre-existing before admission to intensive care
* 4. Patients whose neurological and psychiatric history is unknown prior to resuscitation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients hospitalized in a medical intensive care unit with a neurological disease affecting the central or peripheral nervous system, which is the reason for their hospitalization in an intensive care unit,
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Evaluate the presence at 3 months of discharge from an ICU stay for neurological disease of a post intensive care syndrome defined as a physical symptom | 3 months
  defined by the presence of an MRC (Medical Research Council) score <48/60 (higher score mean better outcome)
Evaluate the presence at 3 months of discharge from an ICU stay for neurological disease of a post intensive care syndrome defined as a cognitive symptom | 3 months
  defined by a MOCA (Montreal Cognitive Assessment) <26/30 (higher score mean better outcome)
Evaluate the presence at 3 months of discharge from an ICU stay for neurological disease of a post intensive care syndrome defined as a psychological symptom | 3 months
  defined by a Hospital Anxiety and Depression Scale (HADS) score A or D > 8 (ranging frome 0 to 21, lower score mean better outcome)
Evaluate the presence at 3 months of discharge from an ICU stay for neurological disease of a post intensive care syndrome defined as a psychological symptom. | 3 months
  defined by an Impact of Events Scale (IESR) > 22 (ranging from 0 to 88, lower score mean better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Clémence Marois, MD, MSc, Principal Investigator — Assisitance Publique des Hôpitaux de Paris
Locations (2):
- France (2):
  - GH Pitié Salpêtrière, Paris
  - CH Saint Anne, Paris

IPD SHARING:
Plan to Share IPD: No